CLINICAL TRIAL: NCT04611347
Title: A Randomized Controlled Trial of Topical Cannabidiol for the Treatment of Thumb Basal Joint Arthritis
Brief Title: Is Topical CBD Effective in Treating Thumb Joint Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Brent DeGeorge, Principal Investigator, University of Virginia
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HSR200147
Record Dates: First submitted 2020-10-02; First posted 2020-11-02 (Actual); Results first posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: CBD; Hand Osteoarthritis

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial with crossover
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Start with CBD (Active Comparator): The study design with be a double-blind, randomized controlled trial with crossover. Treatment will be blinded to the subjects and investigators. Patients will be randomly assigned 2 weeks of the CBD and then crossover to the other condition (Shea butter only ) for 2 additional weeks. Patients will apply the cream at the thumb base twice daily for 1 hour. Subjects will be advised to observe for physiologic changes, skin changes, or other adverse effects.
  Interventions: Drug: CBD; Drug: Shea Butter
- Start with control (Shea butter) (Active Comparator): The study design with be a double-blind, randomized controlled trial with crossover. Treatment will be blinded to the subjects and investigators. Patients will be randomly assigned 2 weeks of Shea butter and then crossover to the other condition (CBD)for 2 additional weeks. Patients will apply the cream at the thumb base twice daily for 1 hour. Subjects will be advised to observe for physiologic changes, skin changes, or other adverse effects.
  Interventions: Drug: CBD; Drug: Shea Butter

INTERVENTIONS:
Drug: CBD — Topical CBD application for thumb basal joint osteoarthritis.
Drug: Shea Butter — Placebo Shae Butter for comparison

SUMMARY:
Rationale: CBD is commonly being used as an over-the-counter treatment for arthritis-related pain, however no clinical trial has been performed to establish efficacy.

Hypothesis: CBD is more effective than placebo for relieving pain and improving patient-reported outcomes for thumb basal joint arthritis.

Study Design: The study design with be a double-blind, randomized controlled trial with crossover. Treatment will be blinded to the subjects and investigators. Patients will be randomly assigned 2 weeks of the CBD or control and then crossover to the other condition for 2 additional weeks. Patients will apply the cream at the thumb base twice daily for 1 hour. Subjects will be advised to observe for physiologic changes, skin changes, or other adverse effects.

DETAILED DESCRIPTION:
Study Population: 40 subjects with presenting with thumb basal joint arthritis over the age of 18 will be recruited from the UVA Hand Center.

Description of Sites/Facilities Enrolling Participants: This will be a single-site study conducted at the UVA Hand Center at the University of Virginia.

Description of Study Intervention: The study design will be a double-blind randomized control trial with crossover. Treatment will be blinded to the subjects and investigators. Patients will be randomly assigned 2 weeks of the case (CBD) or control cream and then crossover to the other cream for 2 more weeks. Patients will apply the topical cream at their thumb basal joint one time daily for 1 hour. The subjects will be advised to observe for physiologic changes, skin changes, or other adverse effects. If mild to serious adverse events are noticed, the creams will be removed immediately and appropriate care and observation will be taken. Each condition will last for 2 weeks and then subjects will be contacted by the study coordinator to facilitate crossover into the other condition. To capture any delayed-onset adverse events, including those related to skin changes that might develop after the drug is discontinued, subjects will attend a follow-up visit seven (7) days following the last dose of investigational cream.

Study Duration: This study will last one year from the beginning of subject recruitment to data analysis.

Participant Duration: Subjects will be enrolled in this study for approximately five (5) weeks from Screening until the final Study Visit.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Provision of signed and dated informed consent form.
2. Stated willingness to comply with all study procedures and availability for the duration of the study.
3. Male or female, aged 18 years or older.
4. Females of childbearing potential must have a negative urine and blood pregnancy test at Screening and a negative urine pregnancy test before study drug is administered. Females must abstain from sex or use a highly effective method of contraception during the period from Screening to administration of study drug and for 30 days after the last dose of study medication. Standard acceptable methods include abstinence or the use of a highly effective method of contraception, including; hormonal contraception, diaphragm, cervical cap, vaginal sponge, condom with spermicide, vasectomy, intrauterine device. If females are of non-child bearing potential, they must be post-menopausal defined as: age > 55 with no menses within the past 12 months, or history of hysterectomy, or history of bilateral oophorectomy, or bilateral tubal ligation.
5. Males must consent to use a medically acceptable method of contraception throughout the entire study period and for 90 days after their last study drug application. They must agree to not donate sperm for 90 days after their last study drug application.
6. Presence of radiographically confirmed diagnosis of thumb basal joint arthritis.

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Subject does not speak English.
2. Severe cardiac, pulmonary, liver and /or renal disease.
3. Coumadin use at time of screening.
4. History of mental illness.
5. Pregnancy or breast feeding at time of screening.
6. Subjects who are incarcerated.
7. History of drug or substance abuse.
8. Pre-existing CBD or hemp based product usage.
9. Subject has had a corticosteroid injection ≤ 3 months prior.
10. Subject has had prior surgery for osteoarthritis treatment.
11. Females who are pregnant, nursing or planning a pregnancy; females of childbearing potential who are unwilling or unable to use an acceptable method of contraception as outlined in this protocol from Screening to the first dose of study medication and for 30 days after the last dose of study medication. Standard acceptable methods include abstinence or the use of a highly effective method of contraception, including; hormonal contraception, diaphragm, cervical cap, vaginal sponge, condom with spermicide, vasectomy, intrauterine device.
12. Any skin disease or condition, including eczema, psoriasis, melanoma, acne or contact dermatitis, scarring, imperfections, lesions, tattoos or discoloration that may affect treatment application, application site assessments, or affect absorption of the study drug.
13. Subjects with ALT/AST >3 times the upper limit of normal at screening.
14. Subjects with history of or active depression or suicide ideation based on Columbia-Suicide Severity Rating Scale (C-SSRS).
15. Subjects taking prescription or non-prescription medication which are substrates of CYP3A4, CYP2C19, CYP2C8, CYP2C9, CYP2C19, CYP1A2 and CYP2B6 within 14 days of the study procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2020-07-28 (Actual); Primary Completion 2021-01-21 (Actual); Study Completion 2022-05-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- First CBD, Then Shea Butter: The study design with be a double-blind, randomized controlled trial with crossover. Treatment will be blinded to the subjects and investigators. Patients will be randomly assigned 2 weeks of the CBD and then crossover to the other condition (Shea butter only ) for 2 additional weeks. Patients will apply the cream at the thumb base twice daily for 1 hour. Subjects will be advised to observe for physiologic changes, skin changes, or other adverse effects.
  CBD: Topical CBD application for thumb basal joint osteoarthritis.
  Shea Butter: Placebo Shae Butter for comparison
- First Shea Butter, the CBD: The study design with be a double-blind, randomized controlled trial with crossover. Treatment will be blinded to the subjects and investigators. Patients will be randomly assigned 2 weeks of Shea butter and then crossover to the other condition (CBD)for 2 additional weeks. Patients will apply the cream at the thumb base twice daily for 1 hour. Subjects will be advised to observe for physiologic changes, skin changes, or other adverse effects.
  CBD: Topical CBD application for thumb basal joint osteoarthritis.
  Shea Butter: Placebo Shae Butter for comparison
Period: Overall Study
Arm/Group | First CBD, Then Shea Butter | First Shea Butter, the CBD
Started | 10 | 8
Completed | 10 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Start With CBD | Start With Control (Shea Butter) | Total
Number analyzed (Participants) | 10 | 8 | 18
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age | 63.6 (13.2) | 64.8 (6.2) | 64.1 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 3 | 2 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White Non-hispanic | 8 | 7 | 15
  African American | 1 | 1 | 2
  Hispanic | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 10 | 8 | 18

OUTCOME MEASURES:

1. Primary Outcome: Change in Hand Strength During Intervention and at Follow-up.
Description: Grip strength, kg.
Time Frame: Change from baseline to 2 weeks
Population: Subjects served as their own control so 18 people completed each intervention.
Measure: Mean (Standard Deviation); unit: KG
Groups:
- CBD Group: The study design with be a double-blind, randomized controlled trial with crossover. Treatment will be blinded to the subjects and investigators. Patients will be randomly assigned 2 weeks of the CBD and then crossover to the other condition (Shea butter only ) for 2 additional weeks. Patients will apply the cream at the thumb base twice daily for 1 hour. Subjects will be advised to observe for physiologic changes, skin changes, or other adverse effects.
  CBD: Topical CBD application for thumb basal joint osteoarthritis. Shea Butter: Placebo Shae Butter for comparison
- Shea Butter Group: The study design with be a double-blind, randomized controlled trial with crossover. Treatment will be blinded to the subjects and investigators. Patients will be randomly assigned 2 weeks of Shea butter and then crossover to the other condition (CBD)for 2 additional weeks. Patients will apply the cream at the thumb base twice daily for 1 hour. Subjects will be advised to observe for physiologic changes, skin changes, or other adverse effects.
  CBD: Topical CBD application for thumb basal joint osteoarthritis. Shea Butter: Placebo Shae Butter for comparison
Arm/Group | CBD Group | Shea Butter Group
Number analyzed (Participants) | 18 | 18
KG | 24 (2.3) | 23 (2.8)

2. Primary Outcome: Change in the PROMIS Upper Extremity Tests During Intervention and at Follow-up.
Description: The Patient Reported Outcome Information System (PROMIS) Upper Extremity Computer Adaptive Test (CAT) is a computerized assessment measuring the physical function of the upper extremity. It is scored using a T-score, and the average is 50 for the U.S. population. In a given PROMIS, a T-score above 50 represents more of the measured variable than the average. For this variable, a T-score above 50 indicates greater physical function than the average population.
Time Frame: Change from baseline to 2 weeks
Population: Subjects served as their own control so 18 people completed each intervention.
Measure: Mean (Standard Deviation); unit: score on a survey
Arm/Group | CBD Group | Shea Butter Group
Number analyzed (Participants) | 18 | 18
score on a survey | 4.2 (1.8) | 38 (1.5)

3. Primary Outcome: Change in Kapandji Score
Description: Kapandji score (ranging 0 to 10) is validated measures in past studies as outcomes for hand disability. The Kapandji score is a tool useful for assessing the opposition of the thumb, based on where on their hand the patient is able to touch with the tip of their thumb. A score of 0 indicates no opposition, a score of 10 indicates maximal opposition.
Time Frame: Change from baseline to 2 weeks
Population: Subjects served as their own control so 18 people completed each intervention.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBD Group | Shea Butter Group
Number analyzed (Participants) | 18 | 18
score on a scale | 9 (0.2) | 9 (0.4)

4. Primary Outcome: Change in Hand Range of Motion
Description: Metacarpal phalangeal (MP) range of motion, passive extension.
Time Frame: Change from baseline to 2 weeks
Population: Subjects served as their own control so 18 people completed each intervention.
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | CBD Group | Shea Butter Group
Number analyzed (Participants) | 18 | 18
degrees | -7.5 (3.9) | -3 (4.2)

5. Secondary Outcome: Rate of Side Effects Using Novel CBD Cream.
Description: Side effects will be assessed at each encounter clinical evaluation by patient report in a Symptom Diary. All side effects thought to be secondary to CBD will be documented.
Time Frame: Change from baseline to 2 weeks
Population: Subjects served as their own control so 18 people completed each intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | CBD Group | Shea Butter Group
Number analyzed (Participants) | 18 | 18
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: AE's were evaluated during the course of the study- 42 days.
Groups:
- CBD Intervention: Time during which subjects were exposed to CBD oil intervention.
- Shea Butter Intervention: Time during which subjects were exposed to Shea Butter intervention.
Arm/Group | CBD Intervention | Shea Butter Intervention
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 0/18 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-04-27): https://cdn.clinicaltrials.gov/large-docs/47/NCT04611347/Prot_SAP_000.pdf
  • Informed Consent Form (2020-05-08): https://cdn.clinicaltrials.gov/large-docs/47/NCT04611347/ICF_001.pdf